CLINICAL TRIAL: NCT01291121
Title: Intravitreal Administration of Ranibizumab Combined With Intravitreous Injection of Expansile Gas and Induction of Posterior Vitreous Detachment in Treatment of Exudative AMD With Posterior VMA: a Pilot, Open Label, Comparative Study
Brief Title: Intravitreal Ranibizumab in Exudative Age-related Macular Degeneration With Posterior Vitreomacular Adhesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2010-0623
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Age related macular degeneration; Intravitreal ranibizumab; Intravitreal expansile gas injection
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- group 1 (Active Comparator): Intravitreal ranibizumab 0.5mg only group
  Interventions: Procedure: Intravitreal expansile gas and ranibizumab injection

INTERVENTIONS:
Procedure: Intravitreal expansile gas and ranibizumab injection — Intravitreal expansile gas (0.3 cc C3F8) and 0.5mg ranibizumab at day 0 Additional 3 monthly loading injection of intravitreal ranibizumab Additional injection of ranibizumab as needed

SUMMARY:
The main objective is to determine the efficacy of intravitreal administration of Ranibizumab combined with intravitreous injection of expansile gas and induction of posterior vitreous detachment on best-corrected visual acuity and ocular coherence tomography (OCT) macular thickness in subjects with neovascular age-related macular degeneration (AMD) with posterior vitreomacular adhesion (VMA).

Secondary objectives are to assess the safety and tolerability of the intravitreal administration of Ranibizumab combined with intravitreous injection of expansile gas.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of severe visual loss in industrialized countries. In recent years, the advent of anti-vascular endothelial growth factor (VEGF) therapies, such as ranibizumab and bevacizumab, has revolutionized neovascular AMD treatment and anti-VEGF has become the standard treatment for choroidal neovascularization (CNV) with a better visual outcome than previous therapies such as photodynamic therapy (PDT). However, one study reported that up to 45% of cases (20 out of 44 eyes) were non-responders showing resistance to anti-VEGF. In these cases, visual acuity did not improve and persistent subretinal fluid remained despite the usual monthly injection of anti-VEGF. A current focus of anti-VEGF treatment is how to determine which eyes will respond to treatment. To date, three genetic studies into the response to treatment for wet AMD have shown that specific genotypes for complement factor H and LOC genes are associated with treatment response. Previous studies have described the relationship between the posterior vitreous and the macula in AMD and have suggested that vitreomacular adhesion (VMA) plays an important role in the development of exudative AMD. In a recent paired eye study, we controlled confounding variables by selecting only patients with unilateral exudative AMD, and showed that eyes with exudative AMD had a significantly higher incidence of posterior VMA than paired normal eyes (P=0.0007). This result indicates that VMA is a possible risk factor for exudative AMD. In another recent study, Mojana and co-workers reported improvement in VA after 25-gauge trans pars plana vitrectomy (TPPV) with hyaloid removal in five patients who had a history of demonstrable VMA and poorly responsive CNV despite aggressive anti-VEGF therapy. We postulated that a subpopulation of exudative AMD cases do not respond to anti-VEGF therapy and that VMA may play a role in this resistance to therapy. The recent results of our study indicate that posterior VMA has a negative effect on visual outcome after intravitreal anti-VEGF treatment for exudative AMD. BCVA did not improve in eyes with posterior VMA despite anti-VEGF treatment. Posterior hyaloid removal by intravitreous injection of expansile gas and induction of posterior vitreous detachment may be considered as a treatment option in patients with VMA who are poor responders to anti-VEGF treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years old
2. Exudative AMD proven by fundus photograph and fluorescein angiography (FA)with VMA proven by OCT
3. Ability to provide written informed consent and comply with study assessments

Exclusion Criteria:

1. Previous anti-VEGF treatment
2. More than three prior treatment with PDT
3. Previous subfoveal focal laser photocoagulation in the study eye
4. Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding day 0
5. Subfoveal fibrosis or atrophy in the study eye
6. History of vitrectomy surgery in the study eye
7. Significant concurrent ocular or macular diseases in the study eye
8. medical Hx such as myocardial infarction, cerebrovascular accident, ischemic cardiomyopathy, non ocular hemorrhage
9. History of Ranibizumab hypersensitivity
10. Presence of active periocular infection and/or endophthalmitis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in visual acuity and central macular thickness at 12 months | 12 months
  Efficacy of intravitreal administration of Ranibizumab combined with intravitreous injection of expansile gas and induction of posterior vitreous detachment on best-corrected visual acuity and ocular coherence tomography (OCT) macular thickness in subjects with exudative age-related macular degeneration (AMD) with posterior vitreomacular adhesion (VMA).
  Visual acuity measurement: logMAR visual acuity with early treatment of diabetic retinopathy study (ETDRS) chart, Macular thickness measurement: OCT

SECONDARY OUTCOMES:
Number of participants with nonocular complications | 12 months
  - Incidence of non ocular complications (thromboembolic events, non ocular hemorrhage, myocardiac infarct etc.)
Number of participants with ocular complications | 12 months
  Incidence of ocular complications (increased intraocular pressure, endophthalmitis, central retinal artery occlusion etc)

CONTACTS AND LOCATIONS:
Overall Officials: Hyuong Jun Koh, Professor, Principal Investigator — Department of ophthalmology, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Klein R, Peto T, Bird A, Vannewkirk MR. The epidemiology of age-related macular degeneration. Am J Ophthalmol. 2004 Mar;137(3):486-95. doi: 10.1016/j.ajo.2003.11.069. PMID 15013873
- [Background] Avery RL, Pieramici DJ, Rabena MD, Castellarin AA, Nasir MA, Giust MJ. Intravitreal bevacizumab (Avastin) for neovascular age-related macular degeneration. Ophthalmology. 2006 Mar;113(3):363-372.e5. doi: 10.1016/j.ophtha.2005.11.019. Epub 2006 Feb 3. PMID 16458968
- [Background] Freeman WR, Falkenstein I. Avastin and new treatments for AMD: where are we? Retina. 2006 Oct;26(8):853-8. doi: 10.1097/01.iae.0000244722.35073.7c. No abstract available. PMID 17031283
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Lux A, Llacer H, Heussen FM, Joussen AM. Non-responders to bevacizumab (Avastin) therapy of choroidal neovascular lesions. Br J Ophthalmol. 2007 Oct;91(10):1318-22. doi: 10.1136/bjo.2006.113902. Epub 2007 May 30. PMID 17537784
- [Background] Brantley MA Jr, Edelstein SL, King JM, Plotzke MR, Apte RS, Kymes SM, Shiels A. Association of complement factor H and LOC387715 genotypes with response of exudative age-related macular degeneration to photodynamic therapy. Eye (Lond). 2009 Mar;23(3):626-31. doi: 10.1038/eye.2008.28. Epub 2008 Feb 22. PMID 18292785
- [Background] Brantley MA Jr, Fang AM, King JM, Tewari A, Kymes SM, Shiels A. Association of complement factor H and LOC387715 genotypes with response of exudative age-related macular degeneration to intravitreal bevacizumab. Ophthalmology. 2007 Dec;114(12):2168-73. doi: 10.1016/j.ophtha.2007.09.008. PMID 18054635
- [Background] Goverdhan SV, Hannan S, Newsom RB, Luff AJ, Griffiths H, Lotery AJ. An analysis of the CFH Y402H genotype in AMD patients and controls from the UK, and response to PDT treatment. Eye (Lond). 2008 Jun;22(6):849-54. doi: 10.1038/sj.eye.6702830. Epub 2007 Apr 27. PMID 17464302
- [Background] Krebs I, Brannath W, Glittenberg C, Zeiler F, Sebag J, Binder S. Posterior vitreomacular adhesion: a potential risk factor for exudative age-related macular degeneration? Am J Ophthalmol. 2007 Nov;144(5):741-746. doi: 10.1016/j.ajo.2007.07.024. Epub 2007 Sep 20. PMID 17884003
- [Background] Lee SJ, Lee CS, Koh HJ. Posterior vitreomacular adhesion and risk of exudative age-related macular degeneration: paired eye study. Am J Ophthalmol. 2009 Apr;147(4):621-626.e1. doi: 10.1016/j.ajo.2008.10.003. Epub 2009 Jan 20. PMID 19159862
- [Background] Mojana F, Cheng L, Bartsch DU, Silva GA, Kozak I, Nigam N, Freeman WR. The role of abnormal vitreomacular adhesion in age-related macular degeneration: spectral optical coherence tomography and surgical results. Am J Ophthalmol. 2008 Aug;146(2):218-227. doi: 10.1016/j.ajo.2008.04.027. Epub 2008 Jun 6. PMID 18538742
- [Background] Ondes F, Yilmaz G, Acar MA, Unlu N, Kocaoglan H, Arsan AK. Role of the vitreous in age-related macular degeneration. Jpn J Ophthalmol. 2000 Jan-Feb;44(1):91-3. doi: 10.1016/s0021-5155(99)00174-4. PMID 10698032
- [Background] Quaranta-El Maftouhi M, Mauget-Faysse M. Anomalous vitreoretinal adhesions in patients with exudative age-related macular degeneration: an OCT study. Eur J Ophthalmol. 2006 Jan-Feb;16(1):134-7. PMID 16496257
- [Background] Lee SJ, Koh HJ. Effects of vitreomacular adhesion on anti-vascular endothelial growth factor treatment for exudative age-related macular degeneration. Ophthalmology. 2011 Jan;118(1):101-10. doi: 10.1016/j.ophtha.2010.04.015. Epub 2010 Aug 3. PMID 20678805